CLINICAL TRIAL: NCT06118073
Title: The Effect of Utilizing Mindfulness Perioperatively on Pain, Opioid Consumption, and Functional Outcomes in Patients With Depression and Anxiety Undergoing Total Knee Arthroplasty: A Randomized Clinical Trial
Brief Title: Effect of Mindfulness on Pain After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YFILL21P.1017
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Total Knee Replacement; Post Operative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total knee replacement with Headspace (Active Comparator): Participants scheduled for primary total knee replacement will be randomized to receive the mindfulness intervention (a smartphone-based mindfulness application).
  Interventions: Other: Headspace; Procedure: Total Knee Replacement
- Total knee replacement without Headspace (Active Comparator): Participants scheduled for primary total knee replacement will not receive the mindfulness intervention.
  Interventions: Procedure: Total Knee Replacement

INTERVENTIONS:
Other: Headspace — Headspace is a smartphone-based application that guides individuals through various mindfulness sessions and has been shown to reduce symptoms of depression, anxiety, and pain. Participants will be required to answer questions regarding anxiety levels and pain for 6 weeks after surgery.
  Arms: Total knee replacement with Headspace
Procedure: Total Knee Replacement — Participant will have total knee replacement surgery

SUMMARY:
This study will be a prospective randomized controlled trial evaluating the effectiveness of using Headspace before and after undergoing total knee replacement surgery. The purpose of this study will be to determine whether using Headspace will help to improve functional outcome scores, decrease pain, and decrease opioid medication use after total knee replacement in patients with depression and/or anxiety. Headspace is a smartphone-based application that guides individuals through various mindfulness sessions and has been shown to reduce symptoms of depression, anxiety, and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary TKA

AND

* Patients with MDD who take medication for MDD and/or Patients with GAD who take medication for GAD
* Patients with MDD and/or Patients with GAD who are being treated for those conditions with psychotherapy by a psychologist or psychiatrist
* Patients with an SF-12 Mental Health Score less than 45.6
* Owning a smartphone (Apple or Android) to be able to download the mindfulness application

Exclusion Criteria:

* Patients undergoing bilateral TKA
* Patients undergoing revision TKA
* Patients with mental health conditions other than MDD and/or GAD
* Patients currently utilizing a mindfulness application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 6 weeks
  postoperative pain will be measured using the Visual Analog Score (VAS)
Participant satisfaction #1 | 6 weeks
  Participant satisfaction will be measured using the 12-Item Short Form (SF-12) questionnaire
Participant satisfaction #2 | 6 weeks
  Participant satisfaction will be measured using the Knee Injury and Osteoarthritis Outcome Score (KOOS Jr.) questionnaire
Participant mental health | 6 weeks
  mental health will be tracked using the Headspace application after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States